CLINICAL TRIAL: NCT06172569
Title: Spartan Stem, World Cup and World Liner Post Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Signature Orthopaedics (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 111-440-100
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Spartan Stem, World Acetabular Cup and World Liner — The Spartan Stem is a wedge-shaped fit and fill design stem with Titanium Plasma Spray(TPS) and Hydroxyapatite (HA) coating.
  The World Acetabular cup is Porous coated and mated with cross-linked polyethylene World Liner

SUMMARY:
The aim of the study is to monitor the performance of the Signature Orthopaedics Spartan Stem, World Acetabular Cup and World Liner as a post-market vigilance and continuous improvement efforts.

DETAILED DESCRIPTION:
The objective of this PMCF Study is to collect data confirming safety, performance and clinical benefits of the Spartan Stem, World Acetabular Cup and the World Liner when used for primary total hip arthroplasty at 2-years follow-up.

The study includes pre-operative, operative, discharge, 1 year post-operative evaluations, where data concerning the performance and safety of the device are gathered.

The revision rate of the components will be monitored as the primary objective, along with pre and post operative measurement of the Oxford Hip Score (OHS), patient-reported outcome measure (PROM) to quantify patient satisfaction.

Radiography analysis will be done to monitor bony response to the implant and qualify the effectiveness of the cementless fixation.

ELIGIBILITY:
Inclusion Criteria:

* patient requires unilateral primary total hip arthroplasty due to non-inflammatory degenerative joint disease (e.g., osteoarthritis, traumatic arthritis, avascular necrosis, dysplasia/DDH)
* patient must be a candidate for use of the products studied, as determined jointly by the surgeon and patient.
* male and non-pregnant female patients aged 18-75
* patients who understand the conditions of the clinical evaluation and are willing to participate for the length of the prescribed follow-up.

Exclusion Criteria:

* patient has active infection or sepsis(treated or untreated) enough to compromise implant stability or postoperative recovery
* patient is a female of child-bearing age and not taking and not taking contraceptive pills
* patient has inadequate bone stock to support the device (e.g. severe osteopenia, family history of severe osteoporosis or osteopenia)
* patient has a known or suspected metal sensitivity
* patient is immuno-suppressed with disease such as AIDS or is receiving high dose of cortico-steroids.
* patient has an emotional or neurological condition that would pre-empt their ability or unwillingness to participate in the clinical evaluation including mental illness, mental retardation or drug abuse
* patient is severely overweight with a BMI>40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Cleveland Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-08 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Spartan Stem, World Acetabular Cup and World Liner Survival Rate | up to 2 years
  The implant survival rate is based on removal of the device for any reason as determined following the Kaplan-Meier method.

SECONDARY OUTCOMES:
Oxford Hip Score (OHS) | up to 2 years
  The OHS is a patient reported outcome measure (PROM) used to quantify patient satisfaction with the treatment. It consists of 12 questions scored 1 to 5 by the patient.

OTHER OUTCOMES:
Radiographic Analysis | up to 2 years.
  Post-operative radiographs of the implant are analysed to identify locations and sizes of radiolucency, indicative of poor fixation. The size, location and progression of radiolucency is monitored. Smaller, non-progressive radiolucencies are preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Piuzzi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No